CLINICAL TRIAL: NCT04873193
Title: Safety and Feasibility of Utilizing a Novel Wearable Device (Leo) for Assessing Respiratory Function in Children With Respiratory Condition - a Pilot Early Phase Clinical Study
Brief Title: Safety and Feasibility of a Novel Device for Assessing Respiratory Function in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OTH-21-02-01
Record Dates: First submitted 2021-04-22; First posted 2021-05-05 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Oscillometry + Pneumotach Procedure with Leo Device measurements (Other): All patients will undergo oscillometry procedure, followed by pneumotach procedure to measure tidal volume in different sitting positions. The Leo device will be worn throughout both procedures to measure the chest electrical impedance and compare against pneumotach measurements.
  Oscillometry and pneumotach are part of standard of care.
  Interventions: Device: Leo device

INTERVENTIONS:
Device: Leo device — Children's respiratory flow and volume measurements will be continuously recorded using the Leo device during oscillometry and pneumotach procedures.
  Other Names: Pneumotachometer (BioPaC systems, Inc., Goleta, CA, USA) connected to anti-bacterial filter and mouth piece.

SUMMARY:
This is an early phase pilot study designed to test the safety and feasibility of using a novel, wireless, wearable device (Leo) for assessing respiratory parameters (lung volume, respiration rate, heart rate and indices related to tidal breathing flow volume loop) in children with respiratory condition (such as asthma).

There is no product currently on the market that is comparable to this novel Leo device

The study consists of a single visit to evaluate the feasibility and safety of using the Leo device on 20 children with clinically stable asthma.

Stable asthmatic children between the age of 3 and 6, inclusive, will be recruited.

There will be no disease-specific intervention, nor changes to the participant's care management program for their asthma.

ELIGIBILITY:
Inclusion Criteria:

* Children aged ≥3 years old and ≤18 years old at time of consent
* Children with a legal guardian able to sign consent for study participation
* Children and caregivers able to read and understand English or Spanish
* Investigator confirmation for diagnosis of clinically stable respiratory condition, such as clinically diagnosed asthma
* Children who are able to follow instructions and complete oscillometry and tidal breathing tasks

Exclusion Criteria:

* - Children <3 and >18 years of age
* Adults (age ≥ 18 years)
* Children with complex medical conditions which may hinder their ability to complete protocol assessments
* Children who do not have a legal guardian to sign informed consent form
* Children with an active skin condition involving the area on the chest wall where the Leo device will be attached. E.g. inflamed and/or infected eczema or other skin conditions involving the anterior chest wall at the time of recruitment
* Child is determined not eligible by the assessment of the PI
* Fever within the 4 weeks prior to enrollment
* Children with any implanted medical devices, E.g. cardiac pacemaker
* Children with any history of known allergic reaction to adhesives or hydrogels, as the ones used with the Leo device
* Children who have taken a bronchodilator in the last 8-24 hours prior to study visit, depending on the type of medication.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Slow vital capacity from Leo device | Baseline
  Agreement and correlation in the lung function parameters derived using the respiratory impedance signals recorded from Leo device, compared to the pneumotachograph (PNT) device. The PNT device readings will be considered the standard of care, and compared against the Leo device to evaluate for device feasibility. This will be done before and after administration of bronchodilator.
Slow vital capacity from PNT device | Baseline
  Agreement and correlation in the lung function parameters derived using the respiratory impedance signals recorded from Leo device, compared to the pneumotachograph (PNT) device. The PNT device readings will be considered the standard of care, and compared against the Leo device to evaluate for device feasibility. This will be done before and after administration of bronchodilator.
Tidal breathing from Leo device | Baseline
  Agreement and correlation in tidal breathing parameters between Leo and the pneumotachograph (PNT) device. The PNT device parameters are considered standard of care, and will be compared against Leo device to evaluate for device feasibility. This will be done before and after administration of bronchodilator.
Tidal breathing from PNT device | Baseline
  Agreement and correlation in tidal breathing parameters between Leo and the pneumotachograph (PNT) device. The PNT device parameters are considered standard of care, and will be compared against Leo device to evaluate for device feasibility. This will be done before and after administration of bronchodilator.

SECONDARY OUTCOMES:
Usability | Baseline
  Clinician, patient and caregiver usability feedback on the use of the Leo device through an IRB approved participant questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Liu, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data only
Supporting Information: Study Protocol, SAP, ICF, CSR